CLINICAL TRIAL: NCT03226639
Title: Predictive Value of Aortic Stiffness on Recurrence of Atrial Fibrillation After Disconnection of Pulmonary Veins.
Brief Title: Predictive Value of Aortic Stiffness on Recurrence of Atrial Fibrillation After Disconnection of Pulmonary Veins (VARIABLE).
Acronym: VARIABLE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL17_0508
Record Dates: First submitted 2017-07-20; First posted 2017-07-24 (Actual); Last update posted 2017-07-24 (Actual); Status verified 2017-07

CONDITIONS: First Ablation of Atrial Fibrillation
Keywords: Atrial Fibrillation; First Ablation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The ablation of atrial fibrillation (FA) by disconnection of pulmonary veins is a burgeoning intervention. It allows a long-term treatment of this arrhythmia with a success rate of about 80%. There are, nevertheless, some recidivism.

Risk factors for recidivism are poorly codified and need further research. Indeed the identification of factors of poor prognosis could lead to not propose this procedure to the patients who present them and at least to inform them of an increased risk of failure.

To date, aortic stiffness has not been studied in the context of assessing the risk factors for FA recurrence after ablation. On a physiopathological level, the aortic stiffness leads to increase left ventricle's post-load. Cardiac remodeling was observed with diastolic dysfunction and increased left atrial size. That may constitute a substrate for FA recurrence.

In the literature, aortic stiffness can be measured in several ways:

1. Measurement of systolo-diastolic variation of the inner diameter of the aorta by scanner or transesophageal Echography (ETO).
2. Measuring of the Pulse Wave Velocity.
3. Measurement of aortic calcifications.

The investigators propose to evaluate the impact of aortic stiffness on the recidivism of FA 6 months after ablation procedure performed in the Croix-Rousse cardiology's department.

ELIGIBILITY:
Inclusion Criteria :

* 18 years old of both sexes,
* Patient carrying a paroxysmal or persistent atrial fibrillation, benefiting from a first procedure of atrial fibrillation's ablation in the in the Croix-Rousse cardiology's department.
* Patient who signed the consent to participate in the study.

Exclusion Criteria :

* Patient carrying a permanent atrial fibrillation
* Patient who're in atrial fibrillation during the ablation
* Atrial fibrillation relapse's history after ablation
* Pregnant and nursing women
* Patients refusal.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient benefiting of a first Atrial Fibrillation's ablation by cryotherapy or radiofrequency within the Service of the Croix Rousse's hospital and having signed a consent for participate in this research.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2016-11 (Actual); Primary Completion 2018-05 (Estimated); Study Completion 2018-05 (Estimated)

PRIMARY OUTCOMES:
Atrial fibrillation recurrences | Month 6
  Atrial fibrillation recurrences after 6 months of ablation by Holter ECG

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Lantelme, Principal Investigator — Hospices Civils de Lyon - Hôpital de la Croix rousse
Locations (1):
- Hospices Civils de Lyon - Hôpital de la Croix Rousse, Lyon, France